CLINICAL TRIAL: NCT03574103
Title: Comparison of Weight Loss Induced by Daily Time-Restricted Feeding Versus Daily Caloric Restriction in Women With Overweight and Obesity
Brief Title: Chronic Effect of Fasting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Adaliene Versiani M. Ferreira, PhD, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Chronic 72774617.6.0000.5149
Record Dates: First submitted 2018-06-19; First posted 2018-06-29 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Overweight and Obesity
Keywords: Obesity; Overweight; Weight loss; Fasting
MeSH Terms: conditions — Overweight; Obesity; Weight Loss; Fasting | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Caloric restriction only (Active Comparator): Participants in this group will receive a eating plan with caloric restriction as dietary weight loss strategy.
  Interventions: Behavioral: Caloric restriction only
- Caloric restriction plus TRF morning (Experimental): Participants in this group will receive a eating plan with caloric and time restriction as dietary weight loss strategy.
  Interventions: Behavioral: Caloric restriction plus TRF morning
- Caloric restriction plus TRF night (Experimental): Participants in this group will receive a eating plan with caloric and time restriction as dietary weight loss strategy.
  Interventions: Behavioral: Caloric restriction plus TRF night

INTERVENTIONS:
Behavioral: Caloric restriction only — Participants in this group will receive a eating plan with caloric restriction (513 to 770 kcal from estimated energy requirements), without restriction in time for feeding, for 8 weeks.
  Arms: Caloric restriction only
Behavioral: Caloric restriction plus TRF morning — Participants in this group will receive a eating plan with caloric restriction (513 to 770 kcal from estimated energy requirements) and 8 hours for eating (from 12 p.m. to 8 p.m.) and 16 hours of fasting, for 8 weeks.
  Arms: Caloric restriction plus TRF morning
Behavioral: Caloric restriction plus TRF night — Participants in this group will receive a eating plan with caloric restriction (513 to 770 kcal from estimated energy requirements) and 8 hours for eating (from 8 a.m. to 4 p.m.) and 16 hours of fasting, for 8 weeks.
  Arms: Caloric restriction plus TRF night

SUMMARY:
The aim of the study is to determine if time-restricted feeding (TRF) is an effective dietary strategy to weight loss after 8 weeks intervention. TRF will be compared with an intervention without restriction in time for feeding. Both strategies will be with caloric restriction.

DETAILED DESCRIPTION:
The participants of the study will be divided in two groups: (1) a group with caloric restriction and without restriction in time for feeding and (2) a group with caloric restriction and restriction in time for feeding. This second group will be subdivided according to the participant's preference: (2.1) first meal at 8 a.m. and last meal at 4 p.m. or (2.2) first meal at 12 p.m. and last meal at 8 p.m. The caloric restriction for all participants will be 513 to 770 kcal from estimated energy requirement.

ELIGIBILITY:
Inclusion Criteria:

* Females;
* Aged between 18 and 59 years old;
* Body mass index equal or greater 25 kg/m²;
* Agree to sign the informed consent.

Exclusion Criteria:

* Any chronic health conditions (e.g. chronic renal failure, autoimmune, heart, and liver disease);
* Thyroid diseases or medications for its treatment;
* Medications known to affect total energy expenditure;
* Use of steroids, immunosuppressants or non-steroidal anti-inflammatory drugs, weight-loss medications, oral hypoglycemic agents or insulin and any medications that influence metabolic and/or inflammatory parameters;
* Previous surgery for weight loss;
* Pregnancy or breast-feeding;
* Smoking;
* Alcohol use (>2 doses/day).

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-07-09 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in body weight | Baseline and weeks 2, 4 and 8
  Body weight will be assessed by mechanical scale

SECONDARY OUTCOMES:
Change in body composition | Baseline and weeks 2, 4 and 8
  Body composition will be assessed by electrical bioimpedance
Change in resting energy expenditure | Baseline and weeks 2, 4 and 8
  Resting energy expenditure will be assessed by indirect calorimetry
Change in self-reported energy intake | Baseline and weeks 2, 4 and 8
  Dietary energy intake will be assessed with 3-days food records
Change in self-reported diet composition | Baseline and weeks 2, 4 and 8
  Dietary macronutrient intake will be assessed with 3-days food records
Change in self-reported intervention adherence | Baseline and weeks 2, 4 and 8
  Adherence will be assessed by daily record of feeding hours
Change in metabolic profile | Baseline and weeks 2, 4 and 8
  Fasting lipids, glucose and free fatty acids
Change in self-reported stress | Baseline and weeks 2, 4 and 8
  Self-reported stress will be assessed by a questionnaire (Perceived Stress Scale). The total of the scale is a sum of scores of 14 questions. Total score can range from zero to 56. The higher the score, the higher the level of stress.
Change in self-reported anxiety | Baseline and weeks 2, 4 and 8
  Self-reported anxiety will be assessed by a questionnaire (Beck Anxiety Inventory). The questionnaire consists of 21 items and the severity of each of them scored from 0 to 3. The degree of anxiety will be classified according to the final score obtained: 0-7 absent or minimum; 8-15 light; 16-25 moderate; 26-63 severe.
Change in self-reported depression | Baseline and weeks 2, 4 and 8
  Self-reported depression will be assessed by a questionnaire (Beck Depression Inventory). The questionnaire consists of 21 items and the severity of each one scored from 0 to 3. The volunteers will be classified according to the score obtained: BDI ≤ 15: without depression; 16 ≤ BDI ≤ 20: dysphoria; BDI> 20: depression.

OTHER OUTCOMES:
High-sensitivity C-reactive protein | Baseline and weeks 2, 4 and 8
  Change will be assessed in blood sample
Insulin | Baseline and weeks 2, 4 and 8
  Change will be assessed in blood sample
Leptin | Baseline and weeks 2, 4 and 8
  Change will be assessed in blood sample
Ghrelin | Baseline and weeks 2, 4 and 8
  Change will be assessed in blood sample
Brain-Derived Neurotrophic Factor (BDNF) | Baseline and weeks 2, 4 and 8
  Change will be assessed in blood sample

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Hospital da Clínicas, Belo Horizonte, Minas Gerais
  - Hospital das Clínicas, Belo Horizonte, Minas Gerais

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717